CLINICAL TRIAL: NCT05153759
Title: EMS Providers' Health Initiative Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Tegan Mansouri, Postdoctoral Associate, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EMS Health
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Shift-work Disorder
Keywords: EMS; Night shift; Nutrition; Insulin resistance; Circadian rhythm
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein (Active Comparator): Consuming a meal composed of 2:1 grams of protein to carbohydrate during the night shift between 7pm-7am
  Interventions: Other: Meal service
- Moderate protein (Placebo Comparator): Consuming a meal composed of 1:1 grams of protein to carbohydrate during the night shift between 7pm-7am
  Interventions: Other: Meal service

INTERVENTIONS:
Other: Meal service — The primary goal is to pilot the feasibility of a meal service intervention in night shift workers

SUMMARY:
This study aims to explore dietary factors that influence glycemic control in night shift EMS providers and to test the feasibility of a dietary intervention among these providers.

DETAILED DESCRIPTION:
This study can be broken down into two phases. Both phases will take place over the course of 3 weeks. During the first week, participants will be scheduled for a single 60-90 minute zoom appointment. During this appointment, informed consent will be obtained, participants will provide health and demographic information, complete several questionnaires, and be familiarized with study protocols. The following week, participants will wear a continuous glucose monitor, actigraph activity monitor, document everything they have to eat and drink, and rate their daily stress levels. Participants will continue this during the final week and will be randomized to consume either a 2:1 or 1:1 protein to carbohydrate ratio during the night shift during this week.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medical service (EMS) provider
* Works night shift only for at least one year
* Provides patient care as primary duty

Exclusion Criteria:

* Diagnosis of a metabolic disease (i.e. diabetes, prediabetes, metabolic syndrome)
* Taking medication to lower blood glucose
* Pregnant or planning to become pregnant
* Diagnosis of kidney disease or impairment
* Allergies or intolerances to study foods
* Digestive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Two weeks
  Daily mean blood glucose
Compliance | Four days
  Percent of participants who adhere to the dietary intervention

SECONDARY OUTCOMES:
Perceived stress | Two weeks
  Daily rating of stress on a scale of one to 10 where 10 is the most stressed the participant has ever been

CONTACTS AND LOCATIONS:
Overall Officials: David Hostler, PhD, Study Chair — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be de-identified and kept in a password protected database (REDcap.com)